CLINICAL TRIAL: NCT01430962
Title: Randomized Controlled Trial Comparing Endobronchial Ultrasound-guided Transbronchial Needle Aspiration (EBUS-TBNA) Performed Under General Anesthesia Versus Conscious Sedation
Brief Title: Endobronchial Ultrasound Guided Transbronchial Needle Aspiration Performed Under General Anesthesia Versus Moderate Sedation
Acronym: EBUS-GA-MS
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Roberto Casal, Assistant Professor of Medicine, Baylor College of Medicine
Other Study IDs: H-27545
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Mediastinal Lymphadenopathies; Mediastinal Masses; Hilar Lymphadenopathies
Keywords: EBUS; mediastinal lymph nodes; mediastinal masses; anesthesia; moderate sedation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- General Anesthesia: Patients will receive Total Intravenous Anesthesia (TIVA) with a combination of Propofol, Ketamine and neuromuscular blockade by anesthesia. Either an LMA or an ETT will be used to secure airway.
- Moderate Sedation: Patients will receive moderate sedation given by the physician performing EBUS with a combination of Versed and Fentanyl per hospital protocol.

SUMMARY:
The purpose of the study is to determine if there are any differences in yield or safety of Endobronchial Ultrasound-guided Transbronchial Needle Aspiration (EBUS-TBNA) (a type of bronchoscopy with biopsy) performed under general anesthesia versus moderate sedation.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18, evaluated by pulmonary physician that require EBUS TBNA for sampling of hilar and/or mediastinal lymphadenopathies or masses
* Patients should be considered eligible to undergo either CS or GA, without contraindications for either one of them, based on the assessment by the pulmonologist who will perform EBUS-TBNA

Exclusion Criteria:

* Pregnancy or breastfeeding women
* Patients deemed poor candidates for general anesthesia by the evaluating physician (e.g., severe coronary artery disease, COPD with FEV1 < 1 liter, uncontrolled hypertension, increased intracranial pressure, reaction to anesthetics)
* Previous reaction to medications routinely used in conscious sedation
* Patients with history of intolerance to either general anesthesia or conscious sedation
* Dementia or other severe cognitive impairment causing inability to understand or consent to the procedure and study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult individuals with suspected mediastinal or hilar lymphadenopathies or masses referred for endobronchial ultrasound-guided biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic Yield | 24 months

SECONDARY OUTCOMES:
Complications rate | 24 months
Time to recovery from anesthesia | 24 months
Tolerance to procedure | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto F. Casal, MD, Principal Investigator — Baylor College of Medicine- Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

REFERENCES:
- [Background] Steinfort DP, Irving LB. Patient satisfaction during endobronchial ultrasound-guided transbronchial needle aspiration performed under conscious sedation. Respir Care. 2010 Jun;55(6):702-6. PMID 20507652
- [Background] Herth FJ, Eberhardt R, Vilmann P, Krasnik M, Ernst A. Real-time endobronchial ultrasound guided transbronchial needle aspiration for sampling mediastinal lymph nodes. Thorax. 2006 Sep;61(9):795-8. doi: 10.1136/thx.2005.047829. Epub 2006 May 31. PMID 16738038
- [Background] Ost DE, Ernst A, Lei X, Feller-Kopman D, Eapen GA, Kovitz KL, Herth FJF, Simoff M; AQuIRE Bronchoscopy Registry. Diagnostic yield of endobronchial ultrasound-guided transbronchial needle aspiration: results of the AQuIRE Bronchoscopy Registry. Chest. 2011 Dec;140(6):1557-1566. doi: 10.1378/chest.10-2914. Epub 2011 Jun 9. PMID 21659432
- [Derived] Casal RF, Lazarus DR, Kuhl K, Nogueras-Gonzalez G, Perusich S, Green LK, Ost DE, Sarkiss M, Jimenez CA, Eapen GA, Morice RC, Cornwell L, Austria S, Sharafkanneh A, Rumbaut RE, Grosu H, Kheradmand F. Randomized trial of endobronchial ultrasound-guided transbronchial needle aspiration under general anesthesia versus moderate sedation. Am J Respir Crit Care Med. 2015 Apr 1;191(7):796-803. doi: 10.1164/rccm.201409-1615OC. PMID 25574801